CLINICAL TRIAL: NCT03738228
Title: Anti PD-L1 (Atezolizumab) as an Immune Primer and Concurrently With Extended Field Chemoradiotherapy for Node Positive Locally Advanced Cervical Cancer
Brief Title: Atezolizumab Before and/or With Chemoradiotherapy in Immune System Activation in Patients With Node Positive Stage IB2, II, IIIB, or IVA Cervical Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2018-02791; NCI-2018-02791 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-GY017 (Other: NRG Oncology); NRG-GY017 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2018-11-08; First posted 2018-11-13 (Actual); Results first posted 2023-07-20 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-10

CONDITIONS: Cervical Adenocarcinoma; Cervical Adenosquamous Carcinoma; Cervical Squamous Cell Carcinoma; Stage IB2 Cervical Cancer AJCC v8; Stage II Cervical Cancer AJCC v8; Stage IIA Cervical Cancer AJCC v8; Stage IIA1 Cervical Cancer AJCC v8; Stage IIA2 Cervical Cancer AJCC v8; Stage IIB Cervical Cancer AJCC v8; Stage IIIB Cervical Cancer AJCC v8; Stage IVA Cervical Cancer AJCC v8
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — atezolizumab; Brachytherapy; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (atezolizumab, standard cisplatin and radiation therapy) (Experimental): Patients receive atezolizumab IV over 30-60 minutes on days -21, 0, and 21 in the absence of disease progression or unacceptable toxicity. Patients also receive standard of care cisplatin chemotherapy IV over 90 minutes on days 0, 7, 14, 21, 28, and 35. Beginning on day 0, patients also receive standard of care radiation therapy once daily (Monday-Friday) for a total of 25 fractions with image guided brachytherapy beginning in week 4, 5, or at the end of radiation therapy.
  Interventions: Drug: Atezolizumab; Radiation: Brachytherapy; Drug: Cisplatin; Radiation: Radiation Therapy
- Arm B (atezolizumab, standard cisplatin and radiation therapy) (Experimental): Patients receive atezolizumab IV over 30-60 minutes on days 0, 21, and 42 in the absence of disease progression or unacceptable toxicity. Patients also receive standard of care cisplatin chemotherapy, radiation therapy, and image guided brachytherapy as in Arm A.
  Interventions: Drug: Atezolizumab; Radiation: Brachytherapy; Drug: Cisplatin; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG 7446; RG-7446; RG7446; RO 5541267; RO-5541267; RO5541267; Tecentriq
Radiation: Brachytherapy — Undergo standard of care image guided brachytherapy
  Other Names: Brachytherapy, NOS; Internal Radiation; Internal Radiation Brachytherapy; Internal Radiation Therapy; Radiation Brachytherapy; Radiation, Internal
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Radiation: Radiation Therapy — Undergo standard of care radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation

SUMMARY:
This phase I trial studies how well atezolizumab before and/or with standard of care chemoradiotherapy works in immune system activation in patients with stage IB2, II, IIIB, or IVA cervical cancer that has spread to the lymph nodes. Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving atezolizumab before and/or with chemoradiotherapy may lower the chance of tumors growing or spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether differences in sequencing of atezolizumab and chemoradiation result in differential immune activation, as determined by clonal expansion of T cell receptor beta (TCRB) repertoires in peripheral blood on day 21.

SECONDARY OBJECTIVES:

I. To investigate the feasibility of administration of the anti PD-L1 antibody (atezolizumab) as an immune primer and concurrent with chemoradiation (CRT) therapy in patients with locally advanced cervical cancer.

II. To determine the nature and degree of toxicity of the anti PD-L1 antibody (atezolizumab) administered as an immune primer and concurrent with chemoradiation (CRT) therapy in patients with locally advanced cervical cancer.

III. To examine the changes in T cell receptor (TCR) clonality, diversity, and frequency in peripheral blood and tissue and correlate this with clinical outcomes, such as the exploratory response assessment on the post-treatment positron emission tomography (PET)-computed tomography (CT) scan and 2-year disease-free survival (DFS).

IV. To assess the predictive value of baseline and on-treatment PD-L1 expression in the tissue in each treatment arm for clinical outcomes using post-treatment PET-CT scan and 2-year DFS as the outcome measures.

EXPLORATORY OBJECTIVES:

I. To explore baseline and on-treatment blood and tissue biomarkers that could predict response to the combination therapy, as correlated to the exploratory clinical endpoint of the week 12 (day 140) PET-CT scan and 2-year DFS.

II. To explore the response assessment on the exploratory and optional post-treatment week 12 (day 140) PET-CT scan and the clinical 2-year disease free survival (DFS).

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive atezolizumab intravenously (IV) over 30-60 minutes on days -21, 0, and 21 in the absence of disease progression or unacceptable toxicity. Patients also receive standard of care cisplatin chemotherapy IV over 90 minutes on days 0, 7, 14, 21, 28, and 35. Beginning on day 0, patients also receive standard of care radiation therapy once daily (Monday-Friday) for a total of 25 fractions with image guided brachytherapy beginning in week 4, 5, or at the end of radiation therapy.

ARM B: Patients receive atezolizumab IV over 30-60 minutes on days 0, 21, and 42 in the absence of disease progression or unacceptable toxicity. Patients also receive standard of care cisplatin chemotherapy, radiation therapy, and image guided brachytherapy as in Arm A.

After completion of study treatment, patients are followed up at 1 and 3 months, and then every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed newly diagnosed advanced cervical cancer (squamous cell carcinoma, adenocarcinoma, and adenosquamous cell carcinoma): Federation of Gynecology and Obstetrics (FIGO) clinical stages IB2/IIA with positive para-aortic nodes, or FIGO clinical stages IIB/IIIB/IVA with positive pelvic or para-aortic lymph nodes (PALN). Pelvic or PALN nodal status confirmed by PET/CT scan or fine needle biopsy or extra peritoneal biopsy or laparoscopic biopsy. The PALN must be inferior to the T12/L1 interspace
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Leukocytes >= 2,500/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL (> 50,000 for patients with hematologic malignancies)
* Hemoglobin >= 8 g/dL (can be transfused with red blood cells pre-study)
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (however, patients with known Gilbert disease who have serum bilirubin level =< 3 x ULN may be enrolled)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x ULN (AST and/or ALT =< 5 x ULN for patients with liver involvement)
* Alkaline phosphatase =< 2.5 x ULN (=< 5 x ULN for patients with documented liver involvement or bone metastases)
* Creatinine clearance =< 1.5 mg/dL to receive weekly cisplatin

  * Patients whose serum creatinine is between 1.5 and 1.9 mg/dL are eligible for cisplatin if there is no hydronephrosis and the estimated creatinine clearance (CCr) is >= 30 ml/min. For the purpose of estimating the CCr, the formula of Cockcroft and Gault for females should be used
* International normalized ratio (INR) and activated partial thromboplastin time (aPTT) =< 1.5 x ULN (this applies only to patients who do not receive therapeutic anticoagulation; patients receiving therapeutic anticoagulation, such as low-molecular-weight heparin or warfarin, should be on a stable dose)
* Patient does not have a known allergy to cisplatin or compounds of similar biologic composition
* Patient is not actively breastfeeding (or has agreed to discontinue breastfeeding before the initiation or protocol therapy)
* Thyroid-stimulating hormone (TSH) within normal limits or normal free T4 in those with abnormal TSH
* Ability to understand and the willingness to sign a written informed consent document
* Patients positive for human immunodeficiency virus (HIV) are allowed on study, but HIV-positive patients must have:

  * A stable regimen of highly active anti-retroviral therapy (HAART)
  * No requirement for concurrent antibiotics or antifungal agents for the prevention of opportunistic infections
  * A CD4 count above 250 cells/mcL and an undetectable HIV viral load on standard polymerase chain reaction (PCR)-based tests

Exclusion Criteria:

* Patients who have received prior radiation therapy to the pelvis or abdominal cavity, PALN radiation, or previous therapy of any kind for this malignancy or pelvic, PALN, or abdominal radiation for any prior malignancy
* Patients with PALN nodal metastasis above the T12/L1 interspace
* Patients who had a radical hysterectomy with positive PALNs are not eligible
* Patients with prior allogeneic bone marrow transplantation or prior solid organ transplantation
* Patients previously treated with systemic anticancer therapy (e.g., chemotherapy, targeted therapy, immunotherapy) within 3 years prior to entering the study
* Treatment with systemic immunosuppressive medications (including, but not limited to, prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 2 weeks prior to cycle 1, day 1

  * Patients who have received acute, low dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea or steroids as CT scan contrast premedication) may be enrolled
  * The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed
* Known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Patients requiring treatment with a RANKL inhibitor (e.g., denosumab) who cannot discontinue it before treatment with atezolizumab
* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis; cirrhosis; fatty liver; and inherited liver disease

  * Patients with past or resolved hepatitis B infection (defined as having a negative hepatitis B surface antigen [HBsAg] test and a positive anti-HBc [antibody to hepatitis B core antigen] antibody test) are eligible
  * Patients positive for hepatitis C virus (HCV) antibody
* History or risk of autoimmune disease, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjogren's syndrome, Bell's palsy, Guillain-Barre syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, or glomerulonephritis

  * Patients with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone are eligible
  * Patients with controlled type 1 diabetes mellitus on a stable insulin regimen or type 2 diabetes mellitus are eligible
  * Patients with eczema, psoriasis, lichen simplex chronicus or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions:

    * Patients with psoriasis must have a baseline ophthalmologic exam to rule out ocular manifestations
    * Rash must cover less than 10% of body surface area (BSA)
    * Disease is well controlled at baseline and only requiring low potency topical steroids (e.g., hydrocortisone 2.5%, hydrocortisone butyrate 0.1%, fluocinolone 0.01%, desonide 0.05%, alclometasone dipropionate 0.05%)
    * No acute exacerbations of underlying condition within the last 12 months (not requiring psoralen plus ultraviolet A radiation [PUVA], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors; high potency or steroids)
* History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest computed tomography (CT) scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Patients with active tuberculosis (TB) are excluded
* Severe infections within 4 weeks prior to cycle 1, day 1, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
* Signs or symptoms of infection within 2 weeks prior to cycle 1, day 1
* Received intravenous (IV) antibiotics within 2 weeks prior to cycle 1, day 1. Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease) are eligible
* Major surgical procedure within 28 days prior to cycle 1, day 1 or anticipation of need for a major surgical procedure during the course of the study
* Administration of a live, attenuated vaccine within 4 weeks before cycle 1, day 1 or anticipation that such a live, attenuated vaccine will be required during the study and up to 5 months after the last dose of atezolizumab

  * Influenza vaccination should be given during influenza season only (approximately October to March). Patients must not receive live, attenuated influenza vaccine within 4 weeks prior to cycle 1, day 1 or at any time during the study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Severe, active co-morbidity defined as follows:

  * Current (within 28 days of cycle 1, day 1) signs and/or symptoms of bowel obstruction
  * Patients who require parental hydration and/or nutrition
  * Patients who require drainage gastrostomy tube
  * Evidence of bleeding diathesis or clinically significant coagulopathy
  * Serious, non-healing or dehiscing wound, active ulcer or untreated bone fracture
  * History of hemoptysis (>= 1/2 teaspoon of bright red blood per episode) within 1 month of study enrollment
* Significant cardiovascular or cerebrovascular disease including:

  * Uncontrolled hypertension (systolic blood pressure [SBP] >= 150; diastolic blood pressure [DBP] >= 90)
  * History of myocardial infarction within 6 months
  * Unstable angina
  * New York Heart Association functional classification II, III or IV
  * Baseline ejection fraction =< 50% as assessed by echocardiogram or multigated acquisition scan (MUGA)
  * Cerebral vascular accident (CVA) or transient ischemic attack (TIA) within 6 months
  * Significant vascular disease (e.g., aortic aneurysm, requiring surgical repair or peripheral arterial thrombosis) within 6 months
* History of abdominal/pelvic or tracheoesophageal fistula or gastrointestinal perforation and/or abscess within 6 months prior to initiation of treatment
* If patients are of child-bearing potential and do not agree to use two forms of birth control then they are ineligible
* Patients who have had a hysterectomy or are planning to have an adjuvant hysterectomy following radiation as part of their cervical cancer treatment are ineligible
* Patients scheduled to be treated with adjuvant consolidation chemotherapy at the conclusion of their standard chemoradiation
* Pregnant women are excluded from this study because radiation therapy has the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with atezolizumab, breastfeeding should be discontinued if the mother is treated with atezolizumab
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for the 5 months (150 days) after the last dose of the study agent. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Patients taking bisphosphonate therapy for symptomatic hypercalcemia. Use of bisphosphonate therapy for other reasons (e.g. osteoporosis) is allowed
* Patients with known primary central nervous system (CNS) malignancy or CNS metastases are excluded
* Patients with a prior known history of vesicovaginal, enterovaginal or colovaginal fistula

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2025-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jyoti S Mayadev, Principal Investigator — NRG Oncology
Locations (16):
- United States (16):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - UC San Diego Moores Cancer Center, La Jolla, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Augusta University Medical Center, Augusta, Georgia
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Mayadev J, Zamarin D, Deng W, Lankes H, O'Cearbhaill R, Aghajanian CA, Schilder R. Anti-PD-L1 (atezolizumab) as an immune primer and concurrently with extended-field chemoradiotherapy for node-positive locally advanced cervical cancer. Int J Gynecol Cancer. 2020 May;30(5):701-704. doi: 10.1136/ijgc-2019-001012. Epub 2019 Dec 22. PMID 31871115

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was activated on 10/26/2018 and closed to accrual on 6/11/2020.
Groups:
- Arm A: Atezolizumab 1200mg day -21, 0, 21. Chemoradiation: Extended field RT weekly Cisplatin x6 doses, Image guided brachytherapy
- Arm B: Atezolizumab 1200mg day 0, 21, 42 Chemoradiation: Extended field RT weekly Cisplatin x6 doses Image Guided Brachytherapy
Period: Overall Study
Arm/Group | Arm A | Arm B
Started | 21 | 19
Completed | 19 | 17
Not Completed | 2 | 2
Not completed — Never received study treatment | 2 | 2

BASELINE CHARACTERISTICS:
Population: Eligible and treated participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 19 | 17 | 36
Age, Customized [Count of Participants; unit: Participants]
  20-29 years | 0 | 3 | 3
  30-39 years | 3 | 2 | 5
  40-49 years | 3 | 8 | 11
  50-59 years | 8 | 3 | 11
  60-69 years | 4 | 1 | 5
  70-79 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 17 | 36
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 1 | 8
  Not Hispanic or Latino | 11 | 16 | 27
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 14 | 13 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Immune Response
Description: The immune response is measured by total T cell receptor beta (TCRB) clonal expansion in peripheral blood at day 21 from baseline using Adaptive Biotechnologies' immunoSEQ platform from Day -21 to Day 21 for group 1 (i.e., Arm A), and from Day 0 to Day 21 for group 2 (i.e., Arm B). The higher number of total TCR clonal expansion indicates better immune response.
Time Frame: Arm A: 42 days from the first dose of Atezolizumab Arm B: 21 days from the first dose of Atezolizumab
Population: Arm A: All eligible participants who received Atezolizumab at Day -21 and Day 0 with TCRB measurements Arm B: All eligible participants who received Atezolizumab at Day 0 with TCRB measurements
Measure: Mean (Standard Deviation); unit: Total number of expanded clones
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 17 | 13
Total number of expanded clones | 132.7 (175.7) | 192.8 (174.4)

2. Secondary Outcome: Percentage of Participants With Dose Limiting Toxicities
Description: A DLT is defined as any drug related adverse effects that occur during treatment period until 30 days after the completion of CRT and meet the criteria as evaluated by NCI CTCAE v.5 unless clearly unrelated to study therapy (e.g., disease progression).
Time Frame: Arm A: 111 days, i.e., from start of the priming dose of atezolizumab until 30 days after the completion of CRT Arm B: 90 days, i.e., from start of CRT until 30 days after the completion of CRT(Chemoradiation therapy).
Population: Eligible participants who have a DLT and have at least one dose of Atezolizumab, or complete protocol therapy until 30 days after the completion of CRT (Chemoradiation Therapy).
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 16 | 14
Percentage of participants | 0 [0 to 17.07] | 21.43 [6.11 to 46.57]

3. Secondary Outcome: Post-treatment 3-month PET/CT Metabolic Response
Description: Percentage of participants with complete post-treatment 3-month PET/CT metabolic response. The post-treatment 3-month PET/CT metabolic response is evaluated based on the ratio of post-treatment week-12 PET-CT SUVmax to base-line PET-CT scan SUV max, and the response will be classified as complete metabolic response for the ratio < 0.34, or classified as partial metabolic response for 0.34 <= the ratio < 0.76, or classified as stable metabolic response for 0.76 <= the ratio < 1.25, or classified as progressive metabolic disease for the ratio >= 1.25.
Time Frame: 3 months after completion of study treatment
Population: Eligible and treated with PET/CT scans at post-treatment 3 months and baseline
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 7 | 12
Percentage of participants | 71.4 [34.1 to 94.7] | 50 [24.5 to 75.5]

4. Secondary Outcome: Adverse Events (Grade 3 or Higher) During Treatment Period as Assessed by Common Terminology Criteria for Adverse Events (CTCAE) Version (v)5
Description: Number of participants with a maximum grade of 3 or higher during treatment period. Adverse events are graded and categorized using CTCAE v5.0.
Time Frame: Arm A: 111 days, i.e., from start of the priming dose of atezolizumab until 30 days after the completion of CRT Arm B 90 days, i.e., from start of CRT until 30 days after the completion of CRT
Population: Eligible and Treated.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 19 | 17
Participants
  Blood and lymphatic system disorders | 4 | 6
  Cardiac Disorders | 1 | 0
  Gastrointestinal Disorders | 2 | 4
  General disorders and administrative site conditions | 1 | 0
  Infections and Infestations | 3 | 2
  Investigations | 2 | 7
  Metabolism and Nutrition Disorders | 0 | 4
  Musculoskeletal and Connective Tissue Disorders | 0 | 2
  Renal and Urinary Disorders | 1 | 0
  Reproductive System and Breast Disorders | 1 | 2

5. Secondary Outcome: T Cell Receptor (TCR) Simpson Clonality
Description: TCR Simpson clonality in peripheral blood is measured at day 21 using Adaptive Biotechnologies' immunoSEQ platform. It quantitates the extent of mono- or oligoclonal dominance within a TCR repertoire by measuring the shape of the clone frequency distribution ranging from 0 to 1, where values approaching 1 indicate a nearly monoclonal population.
Time Frame: Arm A: 42 days from the first dose of Atezolizumab Arm B: 21 days from the first dose of Atezolizumab
Population: Arm A: All eligible participants who received Atezolizumab at Day -21 and Day 0 with TCR measurements Arm B: All eligible participants who received Atezolizumab Day 0 with TCR measurements
Measure: Median (Full Range); unit: Index
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 17 | 13
Index | 0.0505 [0.0102 to 0.2305] | 0.0448 [0.0112 to 0.1355]

6. Secondary Outcome: Pre-treatment PD-L1 Expression
Description: Pre-treatment PD-L1 SP142 positive immune cells in tumor area in formalin-fixed paraffin-embedded (FFPE) biopsy primary tumor tissues
Time Frame: Within 3 days after randomization but before start of study treatment
Population: Eligible and treated without missing PD-L1 measurement
Measure: Median (Full Range); unit: percentage of PDL-1 expression
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 10 | 12
percentage of PDL-1 expression | 0.75 [0 to 8] | 0.5 [0 to 3]

7. Secondary Outcome: Disease-free Survival (DFS) at 2 Years
Description: Percentage of participants who survive disease-free at 2 years, where DFS is defined as the duration of time from study entry to date of first documented recurrence or progression of disease or death, whichever occurs first. Progression is assessed by RECIST 1.1.Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Up to 2 years
Population: Eligible and Treated
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 19 | 17
Percentage of participants | 68.4 [47 to 85.3] | 52.9 [31.1 to 74]

8. Secondary Outcome: T Cell Receptor (TCR) Diversity
Description: TCR diversity in peripheral blood is measured at day 21 by counting the number of unique rearrangements to a common number of T cells using Adaptive Biotechnologies' immunoSEQ platform. A higher TCR diversity indicates a richer TCR repertoire.
Time Frame: Arm A: 42 days from the first dose of Atezolizumab Arm B: 21 days from the first dose of Atezolizumab
Population: Arm A: All eligible participants who received Atezolizumab at Day -21 and Day 0) with TCR measurements Arm B: All eligible participants who received Atezolizumab Day 0 with TCR measurements
Measure: Median (Full Range); unit: number of unique rearrangements
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 17 | 13
number of unique rearrangements | 12118 [4448 to 14740] | 12237 [8366 to 14906]

ADVERSE EVENTS:
Time Frame: Arm A: 111 days, i.e., from start of the priming dose of atezolizumab until 30 days after the completion of CRT Arm B: 90 days, i.e., from start of CRT until 30 days after the completion of CRT. All-Cause Mortality monitored/assessed up to 2 years.
Description: All Adverse Events (AEs) occurring during treatment and up to 30 days after completion of CRT are reported for eligible and treated participants
Arm/Group | Arm A | Arm B
All-Cause Mortality (participants affected / at risk) | 4/19 | 2/17
Serious Adverse Events (participants affected / at risk) | 6/19 | 7/17
Other Adverse Events (participants affected / at risk) | 19/19 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=19) | Arm B (N=17)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Flu Like Symptoms (General disorders) | 1 | 0
Fever (General disorders) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Musculoskeletal And Connective Tissue Disorder - O (Musculoskeletal and connective tissue disorders) | 0 | 1
Vaginal Hemorrhage (Reproductive system and breast disorders) | 1 | 1
Pelvic Pain (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=19) | Arm B (N=17)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Anemia (Blood and lymphatic system disorders) | 10 | 9
Blood And Lymphatic System Disorders - Other (Blood and lymphatic system disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 1 | 0
Cardiac Disorders - Other (Cardiac disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 5 | 4
Hypothyroidism (Endocrine disorders) | 1 | 0
Floaters (Eye disorders) | 3 | 0
Dry Eye (Eye disorders) | 0 | 1
Blurred Vision (Eye disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 13 | 10
Dry Mouth (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 6 | 3
Vomiting (Gastrointestinal disorders) | 7 | 8
Stomach Pain (Gastrointestinal disorders) | 0 | 1
Bloating (Gastrointestinal disorders) | 0 | 2
Rectal Hemorrhage (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 16 | 10
Mucositis Oral (Gastrointestinal disorders) | 1 | 1
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 2
Hemorrhoids (Gastrointestinal disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 2 | 5
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Pain (General disorders) | 1 | 5
Malaise (General disorders) | 0 | 1
Flu Like Symptoms (General disorders) | 1 | 0
Fever (General disorders) | 4 | 2
General Disorders And Administration Site Conditio (General disorders) | 1 | 0
Fatigue (General disorders) | 9 | 9
Edema Limbs (General disorders) | 1 | 2
Localized Edema (General disorders) | 1 | 0
Chills (General disorders) | 2 | 1
Vulval Infection (Infections and infestations) | 0 | 1
Tooth Infection (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 5 | 2
Vaginal Infection (Infections and infestations) | 2 | 0
Skin Infection (Infections and infestations) | 0 | 1
Otitis Externa (Infections and infestations) | 1 | 0
Infections And Infestations - Other (Infections and infestations) | 0 | 1
Upper Respiratory Infection (Infections and infestations) | 1 | 0
Infusion Related Reaction (Injury, poisoning and procedural complications) | 2 | 1
Bruising (Injury, poisoning and procedural complications) | 2 | 0
Weight Loss (Investigations) | 1 | 2
Thyroid Stimulating Hormone Increased (Investigations) | 0 | 1
Platelet Count Decreased (Investigations) | 4 | 7
Neutrophil Count Decreased (Investigations) | 4 | 6
Lymphocyte Count Decreased (Investigations) | 0 | 3
Creatinine Increased (Investigations) | 4 | 0
Lipase Increased (Investigations) | 1 | 0
Blood Bilirubin Increased (Investigations) | 0 | 1
White Blood Cell Decreased (Investigations) | 4 | 6
Aspartate Aminotransferase Increased (Investigations) | 4 | 0
Alkaline Phosphatase Increased (Investigations) | 1 | 1
Alanine Aminotransferase Increased (Investigations) | 4 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 6 | 7
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 6
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 4 | 6
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Anorexia (Metabolism and nutrition disorders) | 5 | 3
Buttock Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 2 | 1
Peripheral Motor Neuropathy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 4 | 3
Paresthesia (Nervous system disorders) | 1 | 1
Dysarthria (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 5 | 4
Insomnia (Psychiatric disorders) | 0 | 2
Depression (Psychiatric disorders) | 2 | 2
Anxiety (Psychiatric disorders) | 3 | 3
Agitation (Psychiatric disorders) | 3 | 1
Urinary Frequency (Renal and urinary disorders) | 2 | 1
Urinary Incontinence (Renal and urinary disorders) | 1 | 0
Urinary Urgency (Renal and urinary disorders) | 3 | 1
Hematuria (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 4 | 1
Cystitis Noninfective (Renal and urinary disorders) | 2 | 0
Chronic Kidney Disease (Renal and urinary disorders) | 1 | 0
Vaginal Perforation (Reproductive system and breast disorders) | 0 | 1
Vaginal Hemorrhage (Reproductive system and breast disorders) | 4 | 5
Vaginal Discharge (Reproductive system and breast disorders) | 3 | 2
Pelvic Pain (Reproductive system and breast disorders) | 3 | 1
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Skin And Subcutaneous Tissue Disorders - Other (Skin and subcutaneous tissue disorders) | 0 | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Vascular Disorders - Other (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Hot Flashes (Vascular disorders) | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-08): https://cdn.clinicaltrials.gov/large-docs/28/NCT03738228/Prot_SAP_000.pdf